CLINICAL TRIAL: NCT03670550
Title: Dynamic ACL Brace: In Vivo Kinematics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Attending surgeon on the project is moving to a different facility
Sponsor: Steadman Philippon Research Institute (Other)
Collaborators: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-31
Record Dates: First submitted 2018-09-06; First posted 2018-09-13 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: ACL Injury; ACL - Anterior Cruciate Ligament Rupture; ACL; ACL - Anterior Cruciate Ligament Deficiency
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Evaluation of knee stability with brace wear. Control is same subject without the brace.
Masking Description: Investigators and participants cannot be blinded as to whether or not the brace is worn.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Knee Brace (Experimental): ACL-reconstruction patients will be issued an Ossur Rebound ACL Brace at the time of enrollment in the study, prior to surgery. They will use this brace throughout their rehab and physical therapy.
  Dynamic X-ray imaging of the knee will take place prior to surgery, and again upon clearance from physical therapy 7-9 months after surgery. The injured knee will be imaged with and without the brace, and the contralateral limb will be imaged for use as a control.
  Interventions: Device: Ossur Rebound ACL Brace

INTERVENTIONS:
Device: Ossur Rebound ACL Brace — ACL-reconstruction patients will be issued an Ossur Rebound ACL Brace at the time of enrollment in the study, prior to surgery. They will use this brace throughout their rehab and physical therapy. The intervention (brace) will be applied only to the surgical limb.

SUMMARY:
The purpose of this study is to evaluate the effect of the Össur Rebound dynamic ACL brace on knee kinematics evaluated using dynamic stereo X-ray (DSX) imaging during functional activities. Brace performance will be evaluated before and after ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral, complete ACL (Anterior Cruciate Ligament) ruptures (must be documented by prior MRI)
* No other concomitant lower extremity injuries and an uninjured contralateral limb
* Acute ACL tears that will be scheduled for ACL reconstruction with Dr. Robert F. LaPrade
* Minimal swelling and pain
* Able and willing to perform the required study activities

Exclusion Criteria:

* Previous surgery or significant injury to either knee
* Relevant surgery, procedure, injury, or condition in the past two years which may affect knee pain or general movement patterns on either side
* Diagnosis of osteoarthritis, rheumatoid conditions, cancers, or other conditions which may affect musculoskeletal health
* Women who are pregnant, or trying/planning to become pregnant during the next 10 months
* Known balance or vestibular disorders
* Persons with a history of significant radiation exposure, whether occupational or medical in nature (Anyone with a history of medical radiation therapy, for cancer or other conditions, is excluded from the study. Those who have an annual occupational radiation exposure greater than 25mSv may not enroll.)
* Persons with a pacemaker, hearing aid, aneurysm clip or artificial heart valve, or other forms of loose metal implants
* Initial MRI exclusion criteria (assessed by clinical MRI obtained as standard of care at time of ACL injury diagnosis): concomitant injury, multi-ligamentous injury, significant meniscal damage
* Allergy or sensitivity to silver or latex
* Adults lacking capacity to consent for themselves

Post-Op Visit Exclusion Criteria

* Participants who do not pass their return-to-sport test within 7-9 months of ACL-Reconstruction surgery will be excluded from the second phase of testing.
* Participants who no longer pass the MRI screening at the time of Phase 2 testing (for example, who have a new loose metal implant), will be excluded from the MRI portion of the testing only.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Dynamic tibiofemoral kinematics during activities of daily living in ACL-deficient knees | <1wk (pre-operative)
  This study will use dynamic stereo x-ray (pulsed bi-plane fluoroscopy) to measure the dynamic movements of the tibiofemoral joint during walking and stair-climbing, focusing on differences in anterior-posterior sliding and internal/external rotation of the tibia relative to femur, between the braced ACL-deficient knee, unbraced ACL-deficient knee, and the contralateral/uninjured knee.
Dynamic tibiofemoral kinematics during sports activities in ACL-reconstructed-knees | 7-9 months (post-operative)
  This study will use dynamic stereo x-ray (pulsed bi-plane fluoroscopy) to measure the dynamic movements of the tibiofemoral joint during dynamic movements and sports activities, focusing on differences in anterior-posterior sliding and internal/external rotation of the tibia relative to femur, between the braced ACL-reconstructed knee, unbraced ACL-reconstructed knee, and contralateral/uninjured knee.

SECONDARY OUTCOMES:
Percent symmetry in 3D motion capture kinematics and kinetics | <1wk; 7-9months
  Whole-body kinematics and ground reaction forces will be calculated to assess joint angle and ground reaction force symmetry between braced and unbraced conditions during activities of daily living (<1wk) and dynamic/sports activities(7-9months post-operatively).
Muscle contribution levels in braced vs unbraced knee | <1wk; 7-9 months
  Electromyography sensors will detect differences in muscle contributions (in major muscles of the lower extremity) between the braced ipsilateral leg, unbraced ipsilateral leg, and contralateral leg during activities of daily living and dynamic sports activities.
Subject Satisfaction | 2 months; 4 months; 7-9 months
  An overall satisfaction score for brace comfort will be obtained from the 'Quebec User Evaluation of Satisfaction with Assistive Technology.'

CONTACTS AND LOCATIONS:
Locations (1):
- Steadman Philippon Research Institute, Vail, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Butler DL, Noyes FR, Grood ES. Ligamentous restraints to anterior-posterior drawer in the human knee. A biomechanical study. J Bone Joint Surg Am. 1980 Mar;62(2):259-70. No abstract available. PMID 7358757
- [Background] Kiapour AM, Murray MM. Basic science of anterior cruciate ligament injury and repair. Bone Joint Res. 2014 Feb 4;3(2):20-31. doi: 10.1302/2046-3758.32.2000241. Print 2014. PMID 24497504
- [Background] Marshall, T., Gelber, J., & Spindler, K. (2016). Postoperative Knee Bracing After Anterior Cruciate Ligament Reconstruction. Operative Techniques in Sports Medicine, 24(1), 55-58. DOI: 10.1053/j.otsm.2015.10.001
- [Background] Cook FF, Tibone JE, Redfern FC. A dynamic analysis of a functional brace for anterior cruciate ligament insufficiency. Am J Sports Med. 1989 Jul-Aug;17(4):519-24. doi: 10.1177/036354658901700412. PMID 2782535
- [Background] Smith SD, Laprade RF, Jansson KS, Aroen A, Wijdicks CA. Functional bracing of ACL injuries: current state and future directions. Knee Surg Sports Traumatol Arthrosc. 2014 May;22(5):1131-41. doi: 10.1007/s00167-013-2514-z. Epub 2013 Apr 27. PMID 23624655
- [Background] Mayr HO, Stueken P, Munch EO, Wolter M, Bernstein A, Suedkamp NP, Stoehr A. Brace or no-brace after ACL graft? Four-year results of a prospective clinical trial. Knee Surg Sports Traumatol Arthrosc. 2014 May;22(5):1156-62. doi: 10.1007/s00167-013-2564-2. Epub 2013 Jun 27. PMID 23807029
- [Background] LaPrade RF, Venderley MB, Dahl KD, Dornan GJ, Turnbull TL. Functional Brace in ACL Surgery: Force Quantification in an In Vivo Study. Orthop J Sports Med. 2017 Jul 6;5(7):2325967117714242. doi: 10.1177/2325967117714242. eCollection 2017 Jul. PMID 28748195